CLINICAL TRIAL: NCT05701384
Title: A Phase II Study for the Evaluation of the Feasibility of Lazertinib 160mg Per Day in Patients With EGFR T790M Mutant Non-small Cell Lung Cancer
Brief Title: Lazertinib 160mg in EGFR T790M NSCLC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Jong-Mu Sun, Professor, Samsung Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SMC 2023-01-17
Record Dates: First submitted 2023-01-17; First posted 2023-01-27 (Actual); Last update posted 2023-01-27 (Actual); Status verified 2023-01

CONDITIONS: Lung Cancer Stage IV; EGFR T790M
MeSH Terms: conditions — Lung Neoplasms | interventions — lazertinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Lazertinib 160mg arm (Experimental)
  Interventions: Drug: Lazertinib

INTERVENTIONS:
Drug: Lazertinib — 160mg po qd

SUMMARY:
The lazertinib is currently approved as 2nd line T790M mutation-positive NSCLC that failed from either 1st or 2nd generation EGFR TKI. The current recommended dosage is 240mg. Based on the promising clinical efficacy of the dose escalation study, this study is designed to evaluatee the clinical efficacy and safety of 160mg lazertinib.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed non-small cell lung cancer
* Patients in a palliative setting who is not applicable for the curative treatment
* EGFR mutation positive patients who received previous 1st or 2nd generation EGFR TKI
* Confirmed EGFR T790M mutation after the previous EGFR TKI
* Available to receive lazertinib either as po or vis levine tube
* Willing to participate clinical trial
* Age over or equal to 19
* ECOG PS 0 to 2

Exclusion Criteria:

* Previously received 3rd generation EGFR TKI
* No clinical benefit is expected based on the investigator's decision
* Uncontrolled symptomatic CNS metastases
* Uncontrolled systemic disease

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 117 (Estimated)
Dates: Start 2023-02-01 (Estimated); Primary Completion 2024-01-31 (Estimated); Study Completion 2025-01-31 (Estimated)

PRIMARY OUTCOMES:
The dose reduction or treatment discontinuation rate | Total 24 months of study period
  Dose who received dosage below 160mg or discontinued due to the adverse event

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, MA, South Korea

IPD SHARING:
Plan to Share IPD: No
The only clinical outcome data will be published